CLINICAL TRIAL: NCT03735979
Title: Multi-arm Optimization of Stroke Thrombolysis (MOST): a Single Blinded, Randomized Controlled Adaptive, Multi-arm, Adjunctive-thrombolysis Efficacy Trial in Ischemic Stroke
Brief Title: Multi-arm Optimization of Stroke Thrombolysis
Acronym: MOST
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Opeolu Makanju Adeoye, Professor and Chair, Department of Emergency Medicine, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-1464; 1U01NS100699-01A1 (NIH)
Record Dates: First submitted 2018-11-07; First posted 2018-11-08 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — argatroban; Eptifibatide

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Argatroban (Experimental): 100µg/kg bolus followed by 3µg/kg per minute for 12 hours
  Interventions: Drug: Argatroban
- Eptifibatide (Experimental): 135µg/kg bolus followed by 0.75µg/kg/min infusion for two hours
  Interventions: Drug: Eptifibatide
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Argatroban — Direct Thrombin Inhibitor - Argatroban is a derivative of arginine that competitively binds to the active site of thrombin thereby preventing fibrin deposition. With a half-life of 30 minutes, argatroban has an immediate anticoagulant effect after IV administration which is rapidly reversed with discontinuation of the drug.
  Arms: Argatroban
Drug: Eptifibatide — GP 2b/3a Receptor Inhibitor - The final step of platelet aggregation is mediated via the GP2b/3a receptor. Eptifibatide was specifically developed to ensure rapid inhibition of platelet aggregation (within 15 minutes), a short half-life (~2 hours) and rapid dissociation from platelets with 50% restoration of platelet function within 2-4 hours of discontinuation.
  Arms: Eptifibatide
Drug: Placebo — IV placebo solution
  Arms: Placebo

SUMMARY:
The primary efficacy objective of the MOST trial is to determine if argatroban (100µg/kg bolus followed by 3µg/kg per minute for 12 hours) or eptifibatide (135µg/kg bolus followed by 0.75µg/kg/min infusion for two hours) results in improved 90-day modified Rankin scores (mRS) as compared with placebo in acute ischemic stroke (AIS) patients treated with standard of care thrombolysis (0.9mg/kg IV rt-PA or 0.25mg/kg IV tenecteplase or TNK) within three hours of symptom onset. Patients may also receive endovascular thrombectomy (ET) per usual care. Time of onset is defined as the last time the patient was last known to be well.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke patients
2. Treated with 0.9mg/kg IV rt-PA or 0.25mg/kg IV TNK within 3 hours of stroke onset or time last known well
3. Age ≥ 18
4. NIHSS score ≥ 6 prior to IV thrombolysis
5. Able to receive assigned study drug within 60 minutes but no later than 75 minutes of initiation of IV thrombolysis

Exclusion Criteria:

1. Known allergy or hypersensitivity to argatroban or eptifibatide
2. Previous stroke in the past 90 days
3. Previous intracranial hemorrhage, neoplasm, subarachnoid hemorrhage, or arterial venous malformation
4. Clinical presentation suggested a subarachnoid hemorrhage, even if initial CT scan was normal
5. Any surgery, or biopsy of parenchymal organ in the past 30 days
6. Trauma with internal injuries or ulcerative wounds in the past 30 days
7. Severe head trauma in the past 90 days
8. Systolic blood pressure persistently >180mmHg post-IV thrombolysis despite antihypertensive intervention
9. Diastolic blood pressure persistently >105mmHg post-IV thrombolysis despite antihypertensive intervention
10. Serious systemic hemorrhage in the past 30 days
11. Known hereditary or acquired hemorrhagic diathesis, coagulation factor deficiency, or oral anticoagulant therapy with INR >1.5
12. Positive urine or serum pregnancy test for women of child bearing potential
13. Glucose <50 or >400 mg/dl
14. Platelets <100,000/mm3
15. Hematocrit <25 %
16. Elevated pre-thrombolysis PTT above laboratory upper limit of normal
17. Creatinine > 4 mg/dl
18. Ongoing renal dialysis, regardless of creatinine
19. Received Low Molecular Weight heparins (such as Dalteparin, Enoxaparin, Tinzaparin) in full dose within the previous 24 hours
20. Abnormal PTT within 48 hours prior to randomization after receiving heparin or a direct thrombin inhibitor (such as bivalirudin, argatroban, dabigatran or lepirudin)
21. Received Factor Xa inhibitors (such as Fondaparinaux, apixaban or rivaroxaban) within the past 48 hours
22. Received glycoprotein IIb/IIIa inhibitors within the past 14 days
23. Pre-existing neurological or psychiatric disease which confounded the neurological or functional evaluations e.g., baseline modified Rankin score >3
24. Other serious, advanced, or terminal illness or any other condition that the investigator felt would pose a significant hazard to the patient if rt-PA, TNK, eptifibatide or argatroban therapy was initiated

    a. Example: known cirrhosis or clinically significant hepatic disease
25. Current participation in another research drug treatment or interventional device trial - Subjects could not start another experimental agent until after 90 days
26. Informed consent from the patient or the legally authorized representative was not or could not be obtained
27. High density lesion consistent with hemorrhage of any degree
28. Large (more than 1/3 of the middle cerebral artery) regions of clear hypodensity on the baseline CT Scan. Sulcal effacement and/or loss of grey-white differentiation alone are not contraindications for treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 514 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Opeolu Adeoye, MD, Principal Investigator — Washington University School of Medicine
Locations (61):
- United States (61):
  - University of Alabama Hospital, Birmingham, Alabama
  - St. Jude Medical Center, Fullerton, California
  - UCSD Health La Jolla, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - UCSD Medical Center - Hillcrest Hospital, San Diego, California
  - San Francisco General Hospital, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - Santa Barbara Cottage Hospital, Santa Barbara, California
  - Yale New Haven Hospital, New Haven, Connecticut
  - Baptist Medical Center Jacksonville, Jacksonville, Florida
  - Mayo Clinic Hospital, Jacksonville, Florida
  - Jackson Memorial Hospital, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tampa General Hospital, Tampa, Florida
  - Grady Memorial Hospital, Atlanta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Javon Bea Hospital - Riverside, Rockford, Illinois
  - Central DuPage Hospital, Winfield, Illinois
  - University of Kansas Hospital, Kansas City, Kansas
  - University of Kentucky Hospital, Lexington, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan University Hospital, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - McLaren Flint, Flint, Michigan
  - Trinity Health Saint Mary's, Grand Rapids, Michigan
  - Fairview Southdale Hospital, Edina, Minnesota
  - University of Minnesota Medical Center Hospital, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - St. Louis University Hospital, St Louis, Missouri
  - Barnes Jewish Hospital, St Louis, Missouri
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - North Shore University Hospital, Manhasset, New York
  - Mount Sinai Beth Israel, New York, New York
  - SUNY Upstate University Hospital, Syracuse, New York
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - Cleveland Clinic Akron General, Akron, Ohio
  - Mercy Health West Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - OSU Wexner Medical Center, Columbus, Ohio
  - St. John Medical Center, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - UPMC Mercy Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Prisma Health Greenville Memorial Hospital, Greenville, South Carolina
  - Vanderbilt University Hospital, Nashville, Tennessee
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann-Texas Medical Center, Houston, Texas
  - South Texas Health System McAllen, McAllen, Texas
  - University of Utah Healthcare, Salt Lake City, Utah
  - UVA Medical Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roy A, Elm J, Ingles JR, Sabagha N, Huang JF, Bentho O, Ranasinghe T, Streib C, Concha M, Khatri P, Vagal A, Wintermark M, Derdeyn CP, Broderick JP, Barreto AD, Adeoye O, Grotta JC. Thrombolysis Alone vs With Argatroban or Eptifibatide: A Prespecified Subgroup Analysis of the MOST Trial. Neurology. 2025 Nov 11;105(9):e214228. doi: 10.1212/WNL.0000000000214228. Epub 2025 Oct 10. PMID 41071964
- [Derived] Rines I, Adeoye O, Barreto AD, Broderick J, Carrozzella J, Chen H, Concha M, Elm J, Grotta JC, Jasne AS, Khatri P, Roy A, Vagal A, Wintermark M, Yoo AJ, Derdeyn CP; MOST Investigators. Intravenous Argatroban or Eptifibatide in Patients Undergoing Mechanical Thrombectomy: A Subgroup Analysis of the MOST Randomized Clinical Trial. JAMA Neurol. 2025 Aug 18;82(10):1004-12. doi: 10.1001/jamaneurol.2025.2794. Online ahead of print. PMID 40824660
- [Derived] Shawkat A, Barreto AD, Broderick JP, Derdeyn CP, Grotta JC, Khatri P, Pizzella S, Rines I, Roy A, Wilson A, Wintermark M, Adeoye OM. Comparison of Local and Centrally Adjudicated Modified Rankin Scale Scores in the MOST Trial. Stroke. 2025 May;56(5):1280-1284. doi: 10.1161/STROKEAHA.124.049825. Epub 2025 Mar 24. PMID 40123511
- [Derived] Adeoye O, Broderick J, Derdeyn CP, Grotta JC, Barsan W, Bentho O, Berry S, Concha M, Davis I, Demel S, Elm J, Gentile N, Graves T, Hoffman M, Huang J, Ingles J, Janis S, Jasne AS, Khatri P, Levine SR, Majjhoo A, Panagos P, Pancioli A, Pizzella S, Ranasinghe T, Sabagha N, Sivakumar S, Streib C, Vagal A, Wilson A, Wintermark M, Yoo AJ, Barreto AD. Adjunctive Intravenous Argatroban or Eptifibatide for Ischemic Stroke. N Engl J Med. 2024 Sep 5;391(9):810-820. doi: 10.1056/NEJMoa2314779. PMID 39231343
- [Derived] Romano JG, Rundek T. Expanding Treatment for Acute Ischemic Stroke beyond Revascularization. N Engl J Med. 2023 Jun 1;388(22):2095-2096. doi: 10.1056/NEJMe2303184. No abstract available. PMID 37256980
- [Derived] Deeds SI, Barreto A, Elm J, Derdeyn CP, Berry S, Khatri P, Moy C, Janis S, Broderick J, Grotta J, Adeoye O. The multiarm optimization of stroke thrombolysis phase 3 acute stroke randomized clinical trial: Rationale and methods. Int J Stroke. 2021 Oct;16(7):873-880. doi: 10.1177/1747493020978345. Epub 2020 Dec 9. PMID 33297893

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Argatroban | Eptifibatide | Placebo
Started | 59 | 227 | 228
Completed (Includes those that died prior to the modified Rankin Scale assessment at 90 days after randomization.) | 56 | 210 | 212
Not Completed | 3 | 17 | 16
Not completed — Lost to Follow-up | 1 | 12 | 14
Not completed — Withdrawal by Subject | 1 | 5 | 2
Not completed — Not due to the above reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Argatroban | Eptifibatide | Placebo | Total
Number analyzed (Participants) | 59 | 227 | 228 | 514
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [60 to 79] | 68 [58 to 79] | 66 [58 to 78] | 67 [58 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 118 | 110 | 256
  Male | 31 | 109 | 118 | 258
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 23 | 14 | 40
  Not Hispanic or Latino | 56 | 203 | 213 | 472
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 7 | 5 | 14
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  Black or African American | 15 | 61 | 53 | 129
  White | 41 | 156 | 170 | 367
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 2 | 0 | 2
NIHSS [Median (Inter-Quartile Range); unit: units on a scale] — National Institute of Health Stroke Scale (NIHSS) scores range from 0 to 42, with higher scores indicating worse neurologic deficit.
  units on a scale | 12 [8 to 18] | 12 [8 to 17] | 11 [7 to 17] | 12 [7 to 17]
IV Thrombolytic [Count of Participants; unit: Participants] — Type of intravenous thrombolytic received within 3 hours after qualifying stroke onset.
  Participants
    recombinant tissue plasminogen activator (rt-PA) | 52 | 157 | 151 | 360
    tenecteplase (TNK) | 7 | 70 | 77 | 154
Stroke Onset to IV Thrombolytic Start [Mean (Standard Deviation); unit: minutes] | 100 (38.5) | 103 (36) | 101 (36.1) | 102 (36.3)
IV Thrombolytic Start to Study Drug Bolus [Mean (Standard Deviation); unit: minutes] | 62 (14.3) | 65 (20.5) | 63 (18.2) | 64 (18.9)
Endovascular Thrombectomy (EVT) received [Count of Participants; unit: Participants] | 27 | 99 | 99 | 225

OUTCOME MEASURES:

1. Primary Outcome: 90-day Utility Weighted Modified Rankin Scores (UW-mRS)
Description: The modified Rankin scale is a 7 point ordinal scale ranging from 0="no symptoms" to 6="death" . For the primary analysis, the scale was analyzed with patient-centered utility weights. We assigned the following utility weights to the seven levels: 10, 9.1,, 7.6, 6.5, 3.3, 0, 0 (with higher scores indicating a better outcome).
Time Frame: 90 days after randomization
Population: Intention-to-treat
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 59 | 227 | 228
score on a scale | 5.2 (3.7) | 6.3 (3.2) | 6.8 (3.0)
Statistical Analysis 1: Comparison: Argatroban vs Placebo; Test type: Superiority; p = 0.002, Bayesian — The "P-value" is the posterior probability that study drug has a higher benefit than control. The a priori threshold for a successful trial is 0.985. The posterior probability that argatroban was better than placebo was 0.002; Primary analysis compared treatment group with placebo, with adjustment for baseline NIHSS score in a Bayesian normal dynamic linear model; Posterior Mean Difference (Final Values) = -1.51, Standard Deviation 0.51 — The posterior mean of study treatment minus placebo
Statistical Analysis 2: Comparison: Eptifibatide vs Placebo; Test type: Superiority; p = 0.04, Bayesian — The P-value is the posterior probability that study drug has a higher benefit than control. The a priori threshold for a successful trial is 0.985. The posterior probability that eptifibitide was better than placebo was 0.04; [statistical method as in outcome 1, analysis 1]; Posterior Mean Difference (Final Values) = -0.5, Standard Deviation 0.29 — The posterior mean of study treatment minus placebo

2. Secondary Outcome: Percentage of Participants With NIHSS Less Than or Equal to 2 at 24 Hours
Description: National Institute of Health Stroke Scale (NIHSS) scores range from 0 to 42, with higher scores indicating worse neurologic deficit. This is a dichotomous analysis with a cutpoint of 0,1,2 defining the event.
Time Frame: 24 hours after randomization
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 59 | 227 | 228
Participants | 14 | 84 | 89

3. Secondary Outcome: Change From Baseline to 24-hour NIHSS
Description: National Institute of Health Stroke Scale (NIHSS) scores range from 0 to 42, with higher scores indicating worse neurologic deficit.
Time Frame: 24 hours after randomization
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 59 | 227 | 228
units on a scale | -5.1 (9.3) | -6.1 (8.4) | -6.3 (6.8)

4. Secondary Outcome: Percentage of Participants With 90-day mRS 0 or 1 (or Return to Their Historical mRS)
Description: The modified Rankin scale (mRS) is a 7 point scale ranging from 0="no symptoms" to 6="death" where lower scores are better outcomes. For patients with a pre-stroke mRS of greater than 0 or 1, these patients had to return to their historical (pre-stroke) value to be counted as a success.
Time Frame: 90 days after randomization
Population: Intention-to-treat sample
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 59 | 227 | 228
Participants | 14 | 82 | 92

5. Secondary Outcome: Percentage of Participants With 90-day mRS 0, 1 or 2 (or Return to Their Historical mRS)
Description: modified Rankin scale is a 7 point scale ranging from 0="no symptoms" to 6="death" where lower scores are better outcomes.
Time Frame: 90 days after randomization
Population: Intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 59 | 227 | 228
Participants | 26 | 126 | 139

6. Secondary Outcome: 90-day mRS
Description: modified Rankin scale is a 7 point ordinal scale ranging from 0="no symptoms at all" to 6="death" where lower scores are better outcomes.
Time Frame: 90 days after randomization
Population: Intention-to-treat
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 59 | 227 | 228
units on a scale | 3 [2 to 5] | 2 [1 to 3] | 2 [1 to 3]

7. Secondary Outcome: 90-day EQ-5D
Description: EuroQol Five-Dimension (EQ-5D) is a measure of health-related quality of life ranging from -0.59 to 1 where 1 is the best possible health state.
Time Frame: 90 days after randomization
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 59 | 227 | 228
score on a scale | 0.6 (0.3) | 0.6 (0.4) | 0.7 (0.3)

8. Secondary Outcome: Pre-thrombectomy Modified TICI Score of 2B.
Description: The modified thrombolysis in cerebral infarction (TICI) score prior to endovascular thrombectomy procedure. The modified pre-thrombectomy TICI score is a 4 point scale with possible values of 0, 1, 2A, and 2B. The values are defined as follows: 0=No flow, 1=Penetration without distal branch filling, 2A=<50% partial reperfusion, and 2B=50%-99% partial reperfusion.
Time Frame: baseline
Population: Only participants that received endovascular thrombectomy are analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 27 | 99 | 99
Participants | 2 | 5 | 6

9. Secondary Outcome: Post-thrombectomy Modified TICI Score of 2B or 3
Description: The modified thrombolysis in cerebral infarction (TICI) score prior to endovascular thrombectomy procedure. The modified post-thrombectomy TICI score is a 5 point scale with possible values of 0, 1, 2A, 2B, 3. The values are defined as follows: 0=No flow, 1=Penetration without distal branch filling, 2A=<50% partial reperfusion, 2B=50%-99% partial reperfusion, and 3=Completed reperfusion
Time Frame: baseline
Population: Only participants that received endovascular thrombectomy are analyzed for this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 27 | 99 | 99
Participants | 22 | 92 | 93

10. Other Pre Specified Outcome: Symptomatic Intracranial Hemorrhage Within 36 Hours (Primary Safety Outcome)
Description: Type 2 parenchymal hemorrhage or a parenchymal hemorrhage remote from the area of infarction with neurologic deterioration (defined as an increase of ≥4 points in the NIHSS score)within 36 hours after randomization.
Time Frame: 36 hours after randomization
Population: Participants that took any amount of study drug (safety sample)
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 54 | 212 | 217
Participants | 2 | 7 | 4

11. Other Pre Specified Outcome: Type 1 or Type 2 Parenchymal Hemorrhage Within 36 Hours (Safety Outcome)
Time Frame: 36 hours after randomization
Population: Participants that took any amount of study drug (safety sample).
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 54 | 212 | 217
Participants | 3 | 18 | 11

12. Other Pre Specified Outcome: Any Intracranial Hemorrhage Within 36 Hours (Safety Outcome)
Description: Symptomatic or asymptomatic intracranial hemorrhage within 36 hours of randomization.
Time Frame: 36 hours after randomization
Population: Participants that took any amount of study drug (safety sample).
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 54 | 212 | 217
Participants | 20 | 51 | 51

13. Other Pre Specified Outcome: Other Major Hemorrhage Other Than Intracranial Hemorrhage Within 7 Days (Safety Outcome)
Description: Other major hemorrhage other than intracranial hemorrhage (resulting in the transfusion of >2 units of packed red cells).
Time Frame: 7 days after randomization
Population: Participants that took any amount of study drug (safety sample).
Measure: Count of Participants; unit: Participants
Arm/Group | Argatroban | Eptifibatide | Placebo
Number analyzed (Participants) | 54 | 212 | 217
Participants | 1 | 2 | 3

ADVERSE EVENTS:
Time Frame: 90 days after randomization
Description: For all-cause mortality, the at-risk population is participants that received any amount of study drug (safety sample). For serious and other adverse events, the at-risk population is all randomized participants (intent to treat sample).
Arm/Group | Argatroban | Eptifibatide | Placebo
All-Cause Mortality (participants affected / at risk) | 13/54 | 25/212 | 17/217
Serious Adverse Events (participants affected / at risk) | 26/59 | 85/227 | 78/228
Other Adverse Events (participants affected / at risk) | 12/59 | 42/227 | 33/228
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Argatroban (N=59) | Eptifibatide (N=227) | Placebo (N=228)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 5 (5) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 2 (2) | 1 (1)
Cardiac arrest (Cardiac disorders) | 3 (3) | 6 (6) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (3)
Chest pain (General disorders) | 2 (2) | 3 (3) | 1 (2)
Corona virus infection (Infections and infestations) | 0 (0) | 4 (4) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 3 (3) | 2 (2)
Subarachnoid haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 5 (5) | 3 (3)
Brain oedema (Nervous system disorders) | 0 (0) | 4 (4) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 3 (3) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 2 (4) | 7 (7) | 5 (6)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 3 (3) | 6 (6)
Ischaemic stroke (Nervous system disorders) | 5 (6) | 7 (8) | 6 (7)
Stroke in evolution (Nervous system disorders) | 2 (2) | 2 (2) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 3 (3) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 5 (5)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7) | 2 (2)
Low frequency SAEs (General disorders) | 16 (21) | 54 (83) | 52 (67) — Any SAE that occurred at an total frequency of less than 1% across all treatment groups
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Argatroban (N=59) | Eptifibatide (N=227) | Placebo (N=228)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 2 (2) | 5 (5) | 3 (3)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 2 (2)
Coronavirus test positive (Infections and infestations) | 0 (0) | 2 (2) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 5 (5) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 2 (2) | 10 (10) | 4 (4)
Haemorrhage intracranial (Nervous system disorders) | 2 (3) | 2 (2) | 2 (2)
Haemorrhagic transformation stroke (Nervous system disorders) | 0 (0) | 2 (2) | 5 (5)
Headache (Nervous system disorders) | 1 (1) | 3 (4) | 5 (5)
Haematoma (Vascular disorders) | 0 (0) | 7 (8) | 4 (4)
Hypotension (Vascular disorders) | 3 (3) | 2 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/79/NCT03735979/Prot_000.pdf
  • Statistical Analysis Plan (2020-10-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT03735979/SAP_001.pdf